CLINICAL TRIAL: NCT06717555
Title: Observational Study on Fetal Growth Restriction Complicated by Early Flowmetric Alterations. ARDEF Adverse or Reverse End Diastolic Flow
Brief Title: Observational Study on Fetal Growth Restriction Complicated by Early Flowmetric Alterations
Acronym: ARDEF
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ARDEF
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Fetal Growth Restriction (FGR)
Keywords: flowmetric alterations; FGR
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to to understand whether the presence of flowmetric alterations in association with early growth retardation (i.e., before 22 weeks gestational age) is associated with worse neonatal and maternal outcomes than intrauterine growth retardation arising later in life.

DETAILED DESCRIPTION:
The study is prospective and retrospective. As far as concerns the retrospective part, patients for whom pregnancy was monitored at the outpatient clinics of the division of Obstetrics and Prenatal Age Medicine will be enrolled. This is necessary to obtain specific information about the complication rate and progression of pregnancies complicated by fetal growth restriction over the past 15 years (2005 to present) followed at our hospital.

In association with this retrospective part, a prospective part of the study will be conducted: all patients will undergo the ultrasound evaluations required by the normal care protocols for pregnancies complicated by growth restriction (controls 2 times a week or three times a week).

In addition to standard ultrasound monitoring, an instrumental assessment will then be performed using the USCOM 1A ® technique, an ultrasound instrument that, by entering the patient's height and weight, is able to calculate, by means of internal algorithms, the diameter of the aortic valve and blood flow through the valve. In addition, the peak pulsatility of the maternal ophthalmic artery, using Doppler ultrasound technique, which appears to be predictive of the risk of developing preeclampsia, will be evaluated.

An echocardiographic acquisition of the fetal heart using STRAIN technique will then be performed in the context of normal ultrasound. Two-dimensional strain is based on the acquisition of a typical myocardial pattern (called finger print), which can be followed during the cardiac cycle. In other words, the software recognizes a small piece of tissue, evaluating its strain. Because of its angle-independence, two-dimensional strain allows global and segmental assessment of myocardial contractility, both longitudinal and radial. In these patients, strain would have the ability to detect a contractility deficit evidenced by a reduction in peak systolic strain and strain rate that, as already demonstrated in the adult, distinguishes areas of increased fibrosis, myocyte loss, and myocardial fiber reorganization (as in the case of disarray). Strain may also be useful in prognostic stratification of heart failure by distinguishing fetuses with particularly impaired contractile capacity. These two additional instrumental assessments, will require no more than 4 minutes more for the complete examination.

Patients will be adequately informed about the purpose and modalities of the study, and informed consent form will be acquired. Patients will be managed according to company protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Single pregnancy
* Ultrasound monitoring and delivery at Policlinico S. Orsola in Bologna, Italy
* Acquisition of informed consent form

Exclusion Criteria:

- Desire to perform Voluntary Interruption of Pregnancy

Ages: 18 Years to 44 Years | Sex: Female
Age Groups: Adult
Study Population: The study group will consist of patients with single pregnancies complicated by intrauterine growth restriction, who access the Pregnancy at Risk Outpatient Clinic, of the Division of Obstetrics and Prenatal Medicine of Policlinico Sant'Orsola to perform the specific diagnostic-care pathway.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Collecting outcomes of pregnancies complicated by growth restriction and early-onset flowmetric alterations | During prenatal ultrasound
  To collect the outcomes of pregnancies complicated by growth restriction and early-onset flowmetric alterations, at prenatal ultrasound, to obtain information useful for counseling these patients (for patients in the retrospective part, from 2005 to the present).
  To analyze the presence of any correlations between different outcomes in this subpopulation of patients with hemodynamic changes (in terms of central and peripheral resistances) of patients and fetuses in pregnancies complicated by placental insufficiency and fetal growth restriction (for patients in the prospective part up to December 2026).

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana Simonazzi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy